CLINICAL TRIAL: NCT03364153
Title: A Phase 2b Randomized, Double-masked, Controlled Trial to Establish the Safety and Efficacy of Zimura™ (Complement C5 Inhibitor) Compared to Sham in Subjects With Autosomal Recessive Stargardt Disease
Brief Title: Zimura Compared to Sham in Patients With Autosomal Recessive Stargardt Disease (STGD1)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OPH2005; 2017-004783-35 (EudraCT Number)
Record Dates: First submitted 2017-12-01; First posted 2017-12-06 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Stargardt's Macular Dystrophy
Keywords: Zimura (previous name); ARC1905; complement factor C5 inhibitor; avacincaptad pegol; STGD1; Izervay; Stargardt Disease 1; Stargardt's Macular Dystrophy
MeSH Terms: conditions — Stargardt Disease | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- avacincaptad pegol (Experimental): Participants will receive avacincaptad pegol monthly for up to 17 Months.
  Interventions: Drug: avacincaptad pegol
- Sham (Sham Comparator): Participants will receive a matching sham monthly for up to 17 Months.
  Interventions: Drug: Sham

INTERVENTIONS:
Drug: avacincaptad pegol — Intravitreal Injection
  Other Names: Zimura (previous name); ARC1905; Izervay
  Arms: avacincaptad pegol
Drug: Sham — Intravitreal Injection
  Arms: Sham

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of avacincaptad pegol intravitreal injection compared to Sham in participants with autosomal recessive Stargardt disease 1 (STGD1).

ELIGIBILITY:
Inclusion Criteria:

* At least two pathogenic mutations of ATP-Binding Cassette (ABC)A4 gene confirmed by a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory
* Best corrected visual acuity in the study eye between 20/20 - 20/200 Snellen equivalent, inclusive

Exclusion Criteria:

* Macular atrophy secondary to any condition other than STGD1 in either eye
* Any prior treatment for STGD1 including gene therapy, stem cell therapy or any prior intravitreal treatment for any indication in either eye
* Participation in an interventional study of a vitamin A derivative </= 3 months prior to screening
* Presence of intraocular inflammation, macular hole, pathologic myopia, epiretinal membrane, evidence of significant vitreo-macular traction, vitreous hemorrhage or aphakia
* Any intraocular surgery or thermal laser within 3 months of trial entry. Any prior thermal laser in the macular region
* Diabetes mellitus
* Hemoglobin A1c (HbA1c) value of >/=6.5%
* Stroke within 12 months of trial entry
* Any major surgical procedure within one month of trial entry or anticipated during the trial
* Any treatment with an investigational agent in the past 60 days for any condition
* Women who are pregnant or nursing
* Known serious allergies to the fluorescein dye used in angiography, povidone iodine, or to the components of the avacincaptad pegol formulation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Rate of change in the area of ellipsoid zone defect | Baseline up to 18 Months
  The area of ellipsoid zone defect will be measured by en face spectral domain-optical coherence tomography (SD-OCT).

SECONDARY OUTCOMES:
Change in best corrected visual acuity | Baseline up to 18 Months
  Best corrected visual acuity (BCVA) will be measured by Early Treatment Diabetic Retinopathy Study [ETDRS] letters chart.
Change in photopic and/or mesopic macular sensitivity | Baseline up to 18 Months
  The photopic and/or mesopic macular sensitivity will be measured by microperimetry (optional assessment).
Rate of change in the area of atrophic lesion (definite decrease in autofluorescence) | Baseline up to 18 Months
  The definite decrease in autofluorescence (DDAF) will be measured by fundus autofluorescence (FAF).
Rate of change in the thickness of the outer nuclear layer | Baseline up to 18 Months
  The thickness of outer nuclear layer will be measured by a horizontal scan through the foveal center using SD-OCT.
Time to persistent vision loss | Baseline up to 18 Months
  Vision loss is defined as BCVA loss >/= 10, 15 or 20 letters from Baseline at two or more consecutive visits through Month 18.
Emergence of at least one new atrophic lesion (DDAF) | Up to 18 Months
  The DDAF will be measured by FAF.
Number of participants with Adverse Events (AEs) | Up to 18 Months
  An AE is defined as any untoward medical occurrence in a participant including unfavorable and unintended signs, symptoms or disease temporally associated with the use of a medicinal product and which does not necessarily have to have a causal relationship to this treatment.
  AEs include illnesses with onset during the trial, or exacerbations of pre-existing illnesses. Exacerbation of pre-existing illness is defined as a significant increase in the severity of the illness as compared to the start of the trial and should be considered when a patient requires new or additional treatment for that illness.
Number of participants with vital sign abnormalities and/or AEs | Up to 18 Months
  Number of participants with potentially clinically significant vital sign values.
Number of participants with ophthalmic abnormalities and/or AEs | Up to 18 Months
  Number of participants with potentially clinically significant ophthalmic variables.
Number of participants with 12-Lead electrocardiogram (ECG) abnormalities and/or AEs | Up to 18 Months
  Number of participants with potentially clinically significant 12-Lead ECG values.
Number of participants with laboratory value abnormalities and/or AEs | Up to 18 Months
  Number of participants with potentially clinically significant laboratory values.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (41):
- United States (17):
  - Retinal Research Institute, Phoenix, Arizona
  - Jules Stein Eye Institute/ David Geffen School of Medicine, Los Angeles, California
  - VitreoRetinal Associates, Gainesville, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Wilmer Eye Institute, Johns Hopkins, Baltimore, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - University of Michigan/Kellogg Eye Center, Ann Arbor, Michigan
  - The Retina Center, Minneapolis, Minnesota
  - Retina Center of NJ, LLC., Bloomfield, New Jersey
  - Casey Eye Institute/Oregon Health & Science University, Portland, Oregon
  - Wills Eye Hospital/Mid Atlantic Retina, Philadelphia, Pennsylvania
  - UPMC Eye Center, Pittsburgh, Pennsylvania
  - Palmetto Retina Center, West Columbia, South Carolina
  - Austin Retina Associates, Austin, Texas
  - Retina Foundation of the Southwest, Dallas, Texas
  - Strategic Clinical Research Group, Willow Park, Texas
  - University of Utah John A. Moran Eye Center, Salt Lake City, Utah
- France (3):
  - Hopital de la Croix-Rousse, Lyon, Auvergne-Rhône-Alpes
  - Creteil University Eye Clinic University Paris EST, Créteil
  - Centre ophtalmologique des Quinzes Vingts, Paris
- Germany (3):
  - University of Bonn, Bonn
  - Augenklinik der LMU München, München
  - University of Tuebingen, Tübingen
- Hungary (5):
  - Budapest Retina Institute, Budapest
  - Semmelweis Egyetem, Budapest
  - University of Debrecen DE KK Szemészeti Klinika, Debrecen
  - Ganglion Medical Center, Pécs
  - Szegedi Tudomanyegyetem, Szent-Gyorgyi Albert Klinikai Kozpont, Szemeszeti Klinika, Szeged
- Israel (5):
  - Rambam Health Care Campus, Haifa
  - Hadassah University Hospital, Jerusalem
  - Rabin Medical Center, Beilinson campus, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Tel-Aviv Sourasky Medical Center, Ichilov Hospital, Tel Aviv
- Italy (5):
  - AOU Policlinico Sant'Orsola Malpighi, U.O. Oftalmologia,, Bologna
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Ospedale San Raffaele, Milan
  - University of Campania Luigi Vanvitelli Eye Clinic, Naples
  - Fondazione Policlinico Tor Vergata, UOSD Patologie Retiniche, Rome
- Institut de la Macula, Barcelona, Spain
- United Kingdom (2):
  - Princess Alexandra Eye Pavillion, Edinburgh
  - Moorfields Eye Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/